CLINICAL TRIAL: NCT00175513
Title: V3: Vancouver-Victoria Valacyclovir Trial for Early Psychosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Dr. William Honer, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C04-0503; FHA: 2005-07; TPD: 094295
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Psychosis
Keywords: Psychosis; early psychosis; first episode psychosis; schizophrenia; schizoaffective; schizophreniform; bipolar disorder; valtrex; valacyclovir.
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Bipolar Disorder | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Valacyclovir (Valtrex)

SUMMARY:
This is an 18 week (2 weeks run-in, 16 weeks double blind) trial, to determine if an antiviral drug, valacyclovir (Valtrex) is helpful in treating the symptoms of psychosis, a form of a mental disorder.

DETAILED DESCRIPTION:
There is evidence that some of the symptoms of psychosis may be related to past infection with common viruses.

Researchers are looking to recruit a total of 100 subjects with evidence in the past, of exposure to at least 1 of 3 viruses. The viruses include herpes type 1 (HSV-1, which causes cold sores of the lip and has affected about 6/10 people in Vancouver), herpes type 2 (HSV-2 which causes genital sores, and has affected less than 1/10 people in Vancouver) and cytomegalovirus (CMV, which causes few symptoms but has affected 8/10 people in Vancouver). People who have been infected with these viruses in the past develop antibodies in the blood. The antibodies can be measured in blood, and are a test of whether or not there was infection in the past, and possibly affecting the symptoms of psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects antipsychotic, mood stabilizing and antidepressant drug treatment must have been stable for at least 3 months, and there is no plan to change the drug treatment during the 4-month phase of the study.
* Subjects must be seropositive for HSV-1, HSV-2 and/or CMV.
* Subjects must achieve a level of understanding and expressive capacity sufficient to communicate adequately with the study coordinator and to participate in cognitive testing.
* Subjects must be able to provide written informed consent.

Exclusion Criteria:

* Females of childbearing age will agree not to become pregnant and will agree to use a medically acceptable method of birth control.
* Inability to participate in cognitive testing due to severe persistent psychosis or other condition.
* Mental handicap.
* Subjects with known hypersensitivity or allergy to valacyclovir or acyclovir.
* Patient taking nontopical antiviral medications with anti-herpes activity on a regular basis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Honer, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Eric Martin Pavilion, Victoria, British Columbia
  - Peace Arch Hospital, White Rock, British Columbia